CLINICAL TRIAL: NCT04607421
Title: AN OPEN-LABEL, MULTICENTER, RANDOMIZED PHASE 3 STUDY OF FIRST-LINE ENCORAFENIB PLUS CETUXIMAB WITH OR WITHOUT CHEMOTHERAPY VERSUS STANDARD OF CARE THERAPY WITH A SAFETY LEAD-IN OF ENCORAFENIB AND CETUXIMAB PLUS CHEMOTHERAPY IN PARTICIPANTS WITH METASTATIC BRAF V600E-MUTANT COLORECTAL CANCER
Brief Title: A Study of Encorafenib Plus Cetuximab With or Without Chemotherapy in People With Previously Untreated Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry); Merck KGaA, Darmstadt, Germany (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4221015; 2023-509405-77-00 (Registry Identifier: CTIS (EU)); BREAKWATER (Other: Pfizer)
Record Dates: First submitted 2020-10-05; First posted 2020-10-29 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Neoplasms
Keywords: Colorectal cancer; Colon cancer; Rectal cancer; Colorectal Neoplasms; Intestinal cancer; Intestinal Neoplasms; Gastrointestinal cancer; Gastrointestinal Neoplasms; Digestive system cancer; Digestive System Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; BREAKWATER Study
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases | interventions — encorafenib; Cetuximab; Oxaliplatin; Irinotecan; Leucovorin; Levoleucovorin; Fluorouracil; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Safety Lead-in Cohort 1 (Experimental): Encorafenib 300 mg orally once daily Cetuximab 500 mg/m2 (120-minute IV infusion) every two weeks Irinotecan 180 mg/m2 (90-minute IV infusion) every two weeks Leucovorin 400 mg/m2 (120-minute IV infusion) every two weeks 5-FU 400 mg/m2 IV bolus, then 5-FU 2400 mg/m2 continuous IV infusion over 46-48 hours every two weeks
  Interventions: Drug: Encorafenib; Drug: Cetuximab; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU
- Safety Lead-in Cohort 2 (Experimental): Encorafenib 300 mg orally once daily Cetuximab 500 mg/m2 (120 minute IV infusion) every two weeks Oxaliplatin 85 mg/m2 (120-minute IV infusion) every two weeks Leucovorin 400 mg/m2 (120-minute IV infusion) every two weeks 5-FU 400 mg/m2 IV bolus, then 5-FU 2400 mg/m2 continuous IV infusion over 46-48 hours every two weeks
  Interventions: Drug: Encorafenib; Drug: Cetuximab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-FU
- Phase 3 Arm A (Experimental): Encorafenib 300 mg orally once daily Cetuximab 500 mg/m2 (120-minute IV infusion) every two weeks
  Interventions: Drug: Encorafenib; Drug: Cetuximab
- Phase 3 Arm B (Experimental): Encorafenib 300 mg orally once daily Cetuximab 500 mg/m2 (120 minute IV infusion) every two weeks Oxaliplatin 85 mg/m2 (120-minute IV infusion) every two weeks Leucovorin 400 mg/m2 (120-minute IV infusion) every two weeks 5-FU 400 mg/m2 IV bolus, then 5-FU 2400 mg/m2 continuous IV infusion over 46-48 hours every two weeks
  Interventions: Drug: Encorafenib; Drug: Cetuximab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-FU
- Phase 3 Arm C (Active Comparator): Every two weeks: Oxaliplatin 85 mg/m2 (120-minute IV infusion) Leucovorin 400 mg/m2 (120-minute IV infusion) 5-FU 400 mg/m2 IV bolus, then 5-FU 2400 mg/m2 continuous IV infusion over 46-48 hours Bevacizumab (optional; given per prescribing instructions) -OR- Every two weeks: Irinotecan 165 mg/m2 (90-minute IV infusion) Oxaliplatin 85 mg/m2 (120-minute IV infusion) Leucovorin 400 mg/m2 (120-minute IV infusion) 5-FU 2400 or 3200 mg/m2 continuous IV infusion over 46 48 hours Bevacizumab (optional; given per prescribing instructions) -OR- Oxaliplatin 130 mg/m2 (120-minute IV infusion) every 3 weeks Capecitabine 1000 mg/m2 oral tablet twice daily on Days 1-14 Bevacizumab (optional; given per prescribing instructions)
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU; Drug: Capecitabine; Drug: Bevacizumab
- Cohort 3 Arm D (Experimental): Encorafenib 300 mg orally once daily Cetuximab 500 mg/m2 (120-minute IV infusion) every two weeks Irinotecan 180 mg/m2 (90-minute IV infusion) every two weeks Leucovorin 400 mg/m2 (120-minute IV infusion) every two weeks 5-FU 400 mg/m2 IV bolus, then 5-FU 2400 mg/m2 continuous IV infusion over 46-48 hours every two weeks
  Interventions: Drug: Encorafenib; Drug: Cetuximab; Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU
- Cohort 3 Arm E (Active Comparator): Irinotecan 180 mg/m2 (90-minute IV infusion) every 2 weeks, Leucovorin 400 mg/m2 (120-minute IV infusion) every 2 weeks, 5-FU 400 mg/m2 IV bolus, then 5-FU 2400 mg/m2 continuous IV infusion over 46-48 hours every two weeks, Bevacizumab (optional; given per prescribing instructions)
  Interventions: Drug: Irinotecan; Drug: Leucovorin; Drug: 5-FU; Drug: Bevacizumab

INTERVENTIONS:
Drug: Encorafenib — 75 mg capsules
  Other Names: Braftovi, PF-07263896, LGX818, ONO-7702
  Arms: Cohort 3 Arm D; Phase 3 Arm A; Phase 3 Arm B; Safety Lead-in Cohort 1; Safety Lead-in Cohort 2
Drug: Cetuximab — Injection for intravenous use 100 mg/vial, 200 mg/vial, or 500 mg/vial
  Other Names: Erbitux
  Arms: Cohort 3 Arm D; Phase 3 Arm A; Phase 3 Arm B; Safety Lead-in Cohort 1; Safety Lead-in Cohort 2
Drug: Oxaliplatin — Powder for solution for intravenous use 50 mg/vial, 100 mg/vial, or 200 mg/vial
  Other Names: Eloxatin
  Arms: Phase 3 Arm B; Phase 3 Arm C; Safety Lead-in Cohort 2
Drug: Irinotecan — Solution for intravenous infusion 40 mg/vial, 100 mg/vial, or 300 mg/vial
  Other Names: Campostar
  Arms: Cohort 3 Arm D; Cohort 3 Arm E; Phase 3 Arm C; Safety Lead-in Cohort 1
Drug: Leucovorin — Injection 50 mg/vial, 100 mg/vial, 200 mg/vial, or 350 mg/vial
  Other Names: Wellcovorin, Fusilev, Khapzory
  Arms: Cohort 3 Arm D; Cohort 3 Arm E; Phase 3 Arm B; Phase 3 Arm C; Safety Lead-in Cohort 1; Safety Lead-in Cohort 2
Drug: 5-FU — Injection for intravenous use 250 mg/vial, 500 mg/vial, or 1000 mg/vial
  Other Names: Fluorouracil
  Arms: Cohort 3 Arm D; Cohort 3 Arm E; Phase 3 Arm B; Phase 3 Arm C; Safety Lead-in Cohort 1; Safety Lead-in Cohort 2
Drug: Capecitabine — 150 mg or 500 mg Tablet
  Other Names: Xeloda
  Arms: Phase 3 Arm C
Drug: Bevacizumab — Optional Injection for intravenous use 100 mg/vial or 400 mg/vial
  Other Names: Zirabev
  Arms: Cohort 3 Arm E; Phase 3 Arm C

SUMMARY:
The purpose of this study is to evaluate two study medicines (encorafenib plus cetuximab) taken alone or together with standard chemotherapy for the potential treatment of colorectal cancer that:

* has spread to other parts of the body (metastatic);
* has a certain type of abnormal gene called "BRAF"; and
* has not received prior treatment.

Participants in this study will receive one of the following study treatments:

* Encorafenib plus cetuximab: These participants will receive encorafenib by mouth at home every day and cetuximab once every two weeks by intravenous (IV) infusion (an injection into the vein) at the study clinic.
* Encorafenib plus cetuximab with chemotherapy: These participants will receive encorafenib and cetuximab in the way described in the bullet above. Additionally, they will receive standard chemotherapy by IV infusion and oral treatment at home.
* Chemotherapy alone: These participants will receive chemotherapy, the standard treatment for this condition, by IV infusion at the study clinics and oral treatment at home.

This study is currently enrolling participants who will receive either encorafenib plus cetuximab with chemotherapy or chemotherapy alone.

The study team will monitor how each participant responds to the study treatment for up to about 3 years.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate whether encorafenib plus cetuximab (EC), alone or in combination with chemotherapy, can improve clinical outcomes relative to current standard of-care chemotherapy in participants with previously untreated BRAF V600E-mutant mCRC. Since encorafenib has not previously been combined with chemotherapy, the tolerability and PK of EC in combination with mFOLFOX6 and in combination with FOLFIRI will be evaluated in separate cohorts in the safety lead-in portion of the trial in order to identify which chemotherapy combination is to be used in the Phase 3 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Safety Lead-In = Male/female ≥ 18 years old
* Phase 3 and Cohort 3: Male/female ≥ 16 years old (where permitted locally)
* Histologically or cytologically confirmed Stage IV CRC that contains BRAF V600E mutation
* Prior systemic treatment in metastatic setting: 0-1 regimens for Safety Lead In; none for Phase 3 and Cohort 3. (Note: Prior adjuvant or neoadjuvant therapy considered metastatic treatment if relapse/metastasis < 6 month from end of adj/neoadjuvant treatment )
* Measurable disease (Phase 3 and Cohort 3)/ Measurable or evaluable disease (Safety Lead-in)
* ECOG PS 0-1
* Adequate organ function

Exclusion Criteria:

* Tumors that are locally confirmed or unknown MSI-H or dMMR unless participant is ineligible to receive immune checkpoint inhibitors due to a pre-existing medical condition
* Active bacterial or viral infections in 2 weeks prior to starting dosing
* Symptomatic brain metastases

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2025-12-08 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
Safety Lead-in Study: Incidence of Dose Limiting Toxicities (DLTs) | After 30 evaluable patients in each cohort complete 1 cycle (up to 28 days), approximately 12 months
  Incidence of dose limiting toxicity defined as any adverse event (AE) or abnormal laboratory value assessed as unrelated to disease, disease progression, intercurrent illness or concomitant medications/therapies occurring during the first 28 days of treatment
Phase 3: Progression free survival, by blinded independent review | Duration of Phase 3, approximately 36 months
  Progression free survival, defined as the time from the date of randomization to the earliest documented disease progression or death due to any cause: encorafenib and cetuximab + mFOLFOX6 (Arm B) vs the Control Arm (Arm C)
Phase 3: Objective response rate by blinded independent review | Duration of Phase 3, approximately 23 months
  Objective response defined as complete response (CR), or partial response (PR) according to RECIST v1.1 based on BICR assessment, from the date of randomization until the date of the first documentation of progression of disease (PD)
Cohort 3: Objective response rate by blinded independent review | Duration of Cohort 3, approximately 15 months.
  Defined as CR, or PR according to RECIST v1.1 based on BICR assessment, from the date of randomization until the date of the first documentation of PD, death or start of new anticancer therapy

SECONDARY OUTCOMES:
Safety Lead-in: Incidence of adverse events | After 30 evaluable patients in each cohort complete 1 cycle (up to 28 days), approximately 12 months
  An adverse event is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship as assessed by CTCAE 4.03
Safety Lead-in: Incidence of abnormal clinical laboratory parameters, abnormal vital signs and abnormal electrocardiograms | After 30 evaluable patients in each cohort complete 1 cycle (up to 28 days), approximately 12 months
  Changes in clinical laboratory parameters, vital signs and electrocardiograms determined clinically significant at the investigator's discretion.
Safety Lead-in: Incidence of dose interruptions, dose modifications and discontinuations due to adverse events | After 30 evaluable patients in each cohort complete 1 cycle (up to 28 days), approximately 12 months
Safety Lead-in: Overall response rate by investigator | After 30 evaluable patients in each cohort complete 1 cycle (up to 28 days), approximately 12 months
  Overall response rate, defined as the proportion of participants who have achieved a confirmed best overall response per RECIST v1.1: encorafenib and cetuximab + mFOLFOX6 or FOLFIRI
Safety Lead-in: Duration of response by Investigator | After 30 evaluable patients in each cohort complete 1 cycle (up to 28 days), approximately 12 months
  Duration of response, defined as the time from the date of first radiographic evidence of response to the earliest documented disease progression per RECIST v1.1, or death due to any cause: encorafenib and cetuximab + mFOLFOX6 or FOLFIRI
Safety Lead-in:Progression free survival by Investigator | After 30 evaluable patients in each cohort complete 1 cycle (up to 28 days), approximately 12 months
  Progression free survival, defined as the time from the first dose to the earliest documented disease progression per RECIST v1.1, or death due to any cause: encorafenib and cetuximab + mFOLFOX6 or FOLFIRI
Safety Lead-in: Time to response by Investigator | After 30 evaluable patients in each cohort complete 1 cycle (up to 28 days), approximately 12 months
  Time to response, defined as the time from first dose to first radiographic evidence of response per RECIST v1.1: encorafenib and cetuximab + mFOLFOX6 or FOLFIRI
Safety Lead-in: Overall survival | After 30 evaluable patients in each cohort complete 1 cycle (up to 28 days), approximately 36 months
  Overall survival defined as the time from the first dose to death due to any cause: encorafenib and cetuximab + mFOLFOX6 or FOLFIRI
Phase 3: Overall survival | Duration of Phase 3, approximately 50 months
  Overall survival, defined as the time from the date of randomization to death due to any cause: encorafenib + cetuximab (Arm A) vs Control Arm (Arm C) and encorafenib + cetuximab +mFOLFOX6 (Arm B) vs Control Arm (Arm C) and encorafenib + cetuximab (Arm A) vs encorafenib + cetuximab +mFOLFOX6 (Arm B)
Phase 3: Overall response rate by Investigator and by blinded independent review | Duration of Phase 3, approximately 36 months
  Overall response rate, defined as the proportion of participants who have achieved a confirmed best overall response per RECIST v1.1: encorafenib + cetuximab (Arm A) vs Control Arm (Arm C) and encorafenib + cetuximab +mFOLFOX6 (Arm B) vs Control Arm (Arm C) and encorafenib + cetuximab (Arm A) vs encorafenib + cetuximab +mFOLFOX6 (Arm B)
Phase 3: Duration of response by Investigator and blinded independent review | Duration of Phase 3, approximately 36 months
  Duration of response, defined as the time from the date of first radiographic evidence of response to the earliest documented disease progression per RECIST v1.1, or death due to any cause: encorafenib + cetuximab (Arm A) vs Control Arm (Arm C) and encorafenib + cetuximab +mFOLFOX6 (Arm B) vs Control Arm (Arm C) and encorafenib + cetuximab (Arm A) vs encorafenib + cetuximab +mFOLFOX6 (Arm B)
Phase 3: Time to response by blinded independent review and by Investigator | Duration of Phase 3, approximately 36 months
  Time to response, defined as the time from first dose to first radiographic evidence of response per RECIST v1.1: encorafenib + cetuximab (Arm A) vs Control Arm (Arm C) and encorafenib + cetuximab +mFOLFOX6 (Arm B) vs Control Arm (Arm C) and encorafenib + cetuximab (Arm A) vs encorafenib + cetuximab +mFOLFOX6 (Arm B)
Phase 3: Progression free survival by Investigator and by blinded independent review | Duration of Phase 3, approximately 36 months
  Progression free survival, defined as the time from the first dose to the earliest documented disease progression per RECIST v1.1, or death due to any cause:: encorafenib + cetuximab (Arm A) vs Control Arm (Arm C) and encorafenib + cetuximab +mFOLFOX6 (Arm B) vs Control Arm (Arm C) and encorafenib + cetuximab (Arm A) vs encorafenib + cetuximab +mFOLFOX6 (Arm B)
Phase 3: Progression free survival 2 by Investigator | Duration of Phase 3, approximately 36 months
  Progression free survival 2, defined as the time from the date of randomization to the second objective disease progression per RECIST v1.1, or death from any cause, whichever occurs first: encorafenib + cetuximab (Arm A) vs Control Arm (Arm C) and encorafenib + cetuximab +mFOLFOX6 (Arm B) vs Control Arm (Arm C) and encorafenib + cetuximab (Arm A) vs encorafenib + cetuximab +mFOLFOX6
Phase 3: Incidence of adverse events | Duration of Phase 3, approximately 36 months
  An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship: encorafenib + cetuximab (Arm A) and encorafenib + cetuximab +mFOLFOX6 (Arm B)
Phase 3: Incidence of abnormal clinical laboratory parameters, abnormal vital signs and abnormal electrocardiograms | Duration of Phase 3, approximately 36 months
  Changes in clinical laboratory parameters, vital signs and electrocardiograms determined clinically significant at the investigator's discretion: encorafenib + cetuximab (Arm A) and encorafenib + cetuximab +mFOLFOX6 (Arm B)
Phase 3: Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30) | Duration of Phase 3, approximately 36 months
  EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Phase 3: Change from Baseline in the EuroQol-5D-5L (EQ-5D-5L) Questionnaire | Duration of Phase 3, approximately 36 months
  The EQ-5D-5L is a standardized measure of health utility that provides a single index value for the participant's health status. It is frequently used for economic evaluations of health care and has been shown to be a valid and reliable instrument, and comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS) that are cognitively undemanding, taking about 2 minutes to complete
Phase 3: Change from Baseline in the Patient Global Impression of Severity (PGIS) | Duration of Phase 3, approximately 36 months
  The PGIS is a single-item questionnaire designed to assess participant's overall impression of disease severity at a given point in time.
Phase 3: Change from Baseline in the Patient Global Impression of Change (PGIC) questionnaires | Duration of Phase 3, approximately 36 months
  The PGIC is a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change in symptoms or quality of life since starting treatment.
Phase 3: Confirm the MSI-status in tumor tissue | Once, pre-treatment
  Summarize MSI-status as determined by retrospective central testing of baseline tumor tissue
Phase 3: To determine the correlation between ctDNA levels, BRAF V600 alterations, and clinical outcome | Predose on Cycle 1 Day 1, 15, Cycle 2 Day 15, Cycle 7 Day 1 and EOT. Arm C sampling on Day 1 of Cycles 1-3, 9 and EOT. EOT is approx 36 months.
  ctDNA levels and BRAF V600 VAF from ctDNA analysis of plasma samples collected at baseline and on treatment
Safety Lead-in: Maximum plasma concentration of encorafenib, LHY746, irinotecan and SN-38 | Cycle 1 Day 1 and Day 15: predose, and 0.75, 1.5, 2.5, 3.5, 5.5 and 7.5 hours after dosing, Cycle 1 Day 3 and Day 17:predose and Cycle 2 through Cycle 6: Day 1 predose. Each cycle is 28 days
Safety Lead-in: Area under the plasma concentration time curve of encorafenib, LHY746, irinotecan and SN-38 | Cycle 1 Day 1 and Day 15: predose, and 0.75, 1.5, 2.5, 3.5, 5.5 and 7.5 hours after dosing, Cycle 1 Day 3 and Day 17:predose and Cycle 2 through Cycle 6: Day 1 predose. Each cycle is 28 days.
Safety Lead-in: Time to maximim plasma concentration time curve of encorafenib, LHY746, irinotecan and SN-38 | Cycle 1 Day 1 and Day 15: predose, and 0.75, 1.5, 2.5, 3.5, 5.5 and 7.5 hours after dosing, Cycle 1 Day 3 and Day 17:predose and Cycle 2 through Cycle 6: Day 1 predose. Each cycle is 28 days
Safety Lead-in: Maximum plasma concentration of encorafenib, LHY746 and oxaliplatin | Cycle 1 Day 1 and Day 15: predose, and 1, 2, 3, 4, 6 and 8 hours after dosing, Cycle 1 Day 3 and Day 17: predose and Cycle 2 through Cycle 6: Day 1 predose. Each cycle is 28 days
Safety Lead-in: Area under the plasma concentration time curve of encorafenib, LHY746 and oxaliplatin | Cycle 1 Day 1 and Day 15: predose, and 1, 2, 3, 4, 6 and 8 hours after dosing, Cycle 1 Day 3 and Day 17: predose and Cycle 2 through Cycle 6: Day 1 predose. Each cycle is 28 days
Safety Lead-in: Clearance of irinotecan, SN-38 and oxaliplatin | Cycle 1 Day 1 and Day 15: predose, and 0.75, 1.5, 2.5, 3.5, 5.5 and 7.5 hours after dosing, Cycle 1 Day 3 and Day 17:predose and Cycle 2 through Cycle 6: Day 1 predose. Each cycle is 28 days
  Changes in exposures of irinotecan and its metabolite (SN-38) on Cycle 1 Day 15 compared to Cycle 1 Day 1 in Cohort 1 (encorafenib and cetuximab + FOLFIRI) Changes in exposures of oxaliplatin on Cycle 1 Day 15 compared to Cycle 1 Day 1 in Cohort 2 (encorafenib and cetuximab + mFOLFOX6)
Safety Lead-in: Time to maximim plasma concentration time curve of encorafenib, LHY746 and oxaliplatin | Cycle 1 Day 1 and Day 15: predose, and 1, 2, 3, 4, 6 and 8 hours after dosing, Cycle 1 Day 3 and Day 17: predose and Cycle 2 through Cycle 6: Day 1 predose. Each cycle is 28 days
Phase 3: Trough concentrations of encorafenib and its metabolite LHY746 | Predose on Cycle 1 through Cycle 6. Each cycle is 28 days
  Trough plasma concentrations in all patients in Arm A and Arm B
Cohort 3: Progression free survival by Investigator and by blinded independent review | Duration of Cohort 3, approximately 21 months
  Progression free survival, defined as the time from the first dose to the earliest documented disease progression per RECIST v1.1, or death due to any cause.
Cohort 3: Overall response rate by investigator | Duration of Cohort 3, approximately 21 months
  Overall response rate, defined as the proportion of participants who have achieved a confirmed best overall response per RECIST v 1.1
Cohort 3: Duration of response by Investigator and by blinded independent review | Duration of Cohort 3, approximately 21 months
  Duration of response, defined as the time from the date of first radiographic evidence of response to the earliest documented disease progression per RECIST v1.1, or death due to any cause
Cohort 3: Time to response by Investigator and by blinded independent review | Duration of Cohort 3, approximately 21 months
  Time to response, defined as the time from the date of randomization to first radiographic evidence of response per RECIST v1.1
Cohort 3: Overall survival | Duration of Cohort 3, approximately 36 months
  Overall survival, defined as the time from the date of randomization to death due to any cause
Cohort 3: Incidence of adverse events | Duration of Cohort 3, approximately 21 months
  An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship: encorafenib + cetuximab (Arm A) and encorafenib + cetuximab +mFOLFOX6 (Arm B)
Cohort 3: Incidence of abnormal clinical laboratory parameters, abnormal vital signs and abnormal electrocardiograms | Duration of Cohort 3, approximately 21 months
  Changes in clinical laboratory parameters, vital signs and electrocardiograms determined clinically significant at the investigator's discretion: encorafenib + cetuximab (Arm A) and encorafenib + cetuximab +mFOLFOX6 (Arm B)
Cohort 3: Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30) | Duration of Cohort 3, approximately 21 months
  EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms.
Cohort 3: Change from Baseline in the EuroQol-5D-5L (EQ-5D-5L) Questionnaire | Duration of Cohort 3, approximately 21 months
  The EQ-5D-5L is a standardized measure of health utility that provides a single index value for the participant's health status. It is frequently used for economic evaluations of health care and has been shown to be a valid and reliable instrument, and comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS) that are cognitively undemanding, taking about 2 minutes to complete
Cohort 3: Change from Baseline in the Patient Global Impression of Severity (PGIS) | Duration of Cohort 3, approximately 21 months
  The PGIS is a single-item questionnaire designed to assess participant's overall impression of disease severity at a given point in time.
Cohort 3: Change from Baseline in the Patient Global Impression of Change (PGIC) questionnaires | Duration of Cohort 3, approximately 21 months
  The PGIC is a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change in symptoms or quality of life since starting treatment.
Cohort 3: Confirm the MSI-status in tumor tissue | Once, pre-treatment
  Summarize MSI-status as determined by retrospective central testing of baseline tumor tissue
Cohort 3: To determine the correlation between ctDNA levels, BRAF V600 alterations, and clinical outcome | Predose on Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 15, Cycle 7 Day 1 and End of Treatment (Duration of Cohort 3, approximately 21 months). Each cycle is 28 days.
  ctDNA levels and BRAF V600 VAF from ctDNA analysis of plasma samples collected at baseline and on treatment
Cohort 3: Trough concentrations of encorafenib and its metabolite LHY746 | Predose on Cycle 1 through Cycle 6. Each cycle is 28 days
  Trough plasma concentrations in all patients in Arm D

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (264):
- United States (60):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona - Scottsdale, Scottsdale, Arizona
  - Keck Hospital of USC, Los Angeles, California
  - LAC & USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center/Investigational Drug Services, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Hospital of USC Pasadena, Pasadena, California
  - Mount Sinai Comprehensive Cancer Center, Aventura, Aventura, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - BRCR Global, Plantation, Florida
  - BRCR Medical Center Inc., Plantation, Florida
  - UChicago Medicine - River East, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - UChicago Medicine at Ingalls - Flossmoor, Flossmoor, Illinois
  - UChicago Medicine Ingalls Memorial, Harvey, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - The University of Chicago Medicine Center for Advanced Care Orland Park, Orland Park, Illinois
  - UChicago Medicine at Ingalls - Tinley Park, Tinley Park, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Barnes- Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Papillion, Nebraska
  - Memorial Sloan Kettering Cancer Center - Basking Ridge, Basking Ridge, New Jersey
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Memorial Sloan Kettering Cancer Center- Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center- Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center - Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - Memorial Sloan Kettering Cancer Center- Nassau, Uniondale, New York
  - Cleveland Clinic Taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Stefanie Spielman Comprehensive Breast Cancer, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio
  - The James Outpatient Care West Campus, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Onc and Heme Care Clinic - Westside, Portland, Oregon
  - Providence St Vincent Medical Center, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The West Clinic. PLLC. dba West Cancer Center, Germantown, Tennessee
  - Henry-Joyce Cancer Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- Argentina (4):
  - Centro Medico San Roque, San Miguel de Tucumán, Tucumán Province
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires
  - Clinica Universitaria Reina Fabiola, Córdoba
  - Hospital Privado Centro Médico de Córdoba, Córdoba
- Australia (11):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - GenesisCare - North Shore, St Leonards, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria
- Belgium (8):
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels, Bruxelles-capitale, Région de
  - Cliniques universitaires Saint-Luc, Brussels, Bruxelles-capitale, Région de
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - AZ Groeninge Campus Kennedylaan, Kortrijk, West-vlaanderen
  - ZNA Middelheim, Antwerp
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
  - GZA Hospitals Campus Sint Augustinus, Wilrijk
- Brazil (8):
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Reichow - Centro de Ensino e Pesquisa, Blumenau, Santa Catarina
  - Clínica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia - Faculdade de Medicina do ABC, Santo André, São Paulo
  - FUNDAÇÃO DO ABC - Faculdade de Medicina do ABC - Centro de Estudos e Pesquisas de Hematologia e Onco, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
- Bulgaria (7):
  - MHAT Uni Hospital OOD, Panagyurishte, Pazardzhik
  - MHAT "Dr. Tota Venkova" AD, Gabrovo
  - MHAT Central Onco Hospital OOD, Plovdiv
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Medical Center Nadezhda Clinical EOOD, Sofia
  - Acibadem City Clinic MHAT Tokuda, Sofia
  - University Multiprofile Hospital for Active Treatment Sofiamed, Sofia
- Canada (5):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program, London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- China (21):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - Shandong province cancer hospital, Jinan, Shandong
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Sichuan Province Cancer Hospital, Chengdu, Sichuan
  - Yunnan Cancer Hospital(The Third Affiliated Hospital of Kunming Medical University), Kunming, Yunnan
  - The second Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Union Medical Center, Tianjin
- Czechia (5):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Hradec Králové
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Bulovka, Prague
- Denmark (6):
  - Aalborg Universitetshospital, Syd, Aalborg, North Denmark
  - Vejle Hospital-Sygehus Lillebaelt, Vejle, Region Syddanmark
  - Vejle Sygehus, Vejle, Region Syddanmark
  - Rigshospitalet, Copenhagen
  - Herlev and Gentofte Hospital, Herlev
  - Odense University Hospital, Odense C
- Finland (6):
  - Docrates Syöpäsairaala, Helsinki, Uusimaa
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Satakunnan Keskussairaala, Pori
  - Tampereen yliopistollinen sairaala, Tampere
  - Turku University Hospital, Turku
- Germany (12):
  - Muenchen Klinik Neuperlach, Klinik fuer Haematologie und Onkologie, Munich, Bavaria
  - Institut für Klinisch Onkologische Forschung, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Onkologische Schwerpunktpraxis Kurfuerstendamm, Berlin
  - HELIOS Klinikum Berlin Buch GmbH, Berlin
  - Radiologie Berlin, Charlottenburg
  - Technische Universität Dresden, Medizinische Fakultät Carl Gustav Carus, Dresden
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Facharztzentrum Eppendorf, Hamburg
  - ZytoService Deutschland GmbH, Standort-Hamburg-Jenfeld, Hamburg
  - Radiologie im Israelitischen Krankenhaus, Hamburg
- India (7):
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Bhakti Vedanta Hospital and Research Institute, Thane, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
  - R K Birla Cancer Center, SMS Hospital, Jaipur, Rajasthan
  - Sawai Man Singh Medical College Hospital (SMS Hospital), Jaipur, Rajasthan
- Italy (10):
  - Azienda Ospedaliera Universitaria di Cagliari - Presidio Policlinico Universitario "D.Casula", Monserrato (CA), Cagliari
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milano
  - Fondazione del Piemonte per l'Oncologia - Istituto di Candiolo IRCCS, Candiolo, Torino
  - Azienda Ospedaliero Universitaria San Luigi Gonzaga, Orbassano, Torino
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Azienda Ospedaliera Universitaria dell'Università "Luigi Vanvitelli" di Napoli, Napoli
  - IRCCS Istituto Oncologico Veneto (IOV), Padua
  - Azienda USL - IRCCS di Reggio Emilia - Arcispedale Santa Maria Nuova, Reggio Emilia
- Japan (19):
  - Chiba cancer center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Aichi Cancer Center Hospital, Nagoya, Nagoya, Aichi
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Saitama Prefectural Cancer Center, Ina-machi, Saitama
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research, Osaka
  - Keio university hospital, Tokyo
- Mexico (2):
  - Accelerium, S. de R.L. de C.V., Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL), Amsterdam, North Holland
  - Universitair Medisch Centrum Utrecht, Utrecht
- Auckland City Hospital, Auckland, New Zealand
- Norway (4):
  - St. Olavs hospital, Trondheim, Sør-trøndelag
  - Sørlandet Sykehus Kristiansand, Kristiansand, Vest-agder
  - Oslo universitetssykehus, Radiumhospitalet, Oslo
  - Oslo Universitetssykehus Ullevål, Oslo
- Poland (5):
  - Przychodnia Lekarska KOMED, Konin, Greater Poland Voivodeship
  - Szpital Specjalistyczny W Brzozowie, Podkarpacki Osrodek Onkologiczny Im.Ks.B.Markiewicza, Brzozów
  - Wojewodzki Szpital Specjalistyczny Nr 4 w Bytomiu Oddzial Onkologii, Bytom
  - COPERNICUS PL sp. z. o. o. Wojewodzkie Centrum Onkologii w Gdansku Ambulatoryjna, Gdansk
  - COPERNICUS Podmiot Leczniczy Sp. z o.o. Wojewodzkie Centrum Onkologii, Gdansk
- Russia (11):
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - GBUZ, Chelyabinsk
  - Kaluga Regional Clinical Oncology Center, Kaluga
  - FSAEI HE I.M Sechenov First MSMU MoH Russia (Sechenovskiy University),, Moscow
  - BHI of Omsk Region "Clinical Oncology Dispensary", Omsk
  - LLC "Medicina Severnoy Stolitsy", Saint Petersburg
  - LLC "Severo-Zapadny Medical Center", Saint Petersburg
  - Private Healthcare Institution "Clinical Hospital "RZD-Medicine" of St. Petersburg, Saint Petersburg
  - LLC "EuroCityClinic", Saint Petersburg
  - FSBI "Russian Scientific Center For Radiology and Surgical Technologies n.a. Academician A.M. Granov, Saint Petersburg
  - SHI YR Regional Clinical Oncology Hospital, Yaroslavl
- Slovakia (2):
  - Narodny Onkologicky Ustav, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
- South Africa (3):
  - Cancercare Rondebosch Oncology, Rondebosch, CAPE TOWN
  - Cancercare Langenhoven Drive Oncology Centre, Port Elizabeth, Eastern Cape
  - Wits Health Consortium (Pty) Ltd, Johannesburg
- South Korea (10):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu, Taegu-kwangyǒkshi
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (12):
  - Complejo Hospitalario Universitario Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital General Universitario de Elche, Elche, Alicante
  - ICO L'Hospitalet (Hospital Duran i Reynals), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (4):
  - Karolinska Universitetssjukhuset Solna, Solna, Stockholms LÄN [se-01]
  - Akademiska sjukhuset, Uppsala, Uppsala LÄN [se-03]
  - Norrlands universitetssjukhus, Umeå, Västerbottens LÄN [se-24]
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands LÄN [se14]
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Ukraine (4):
  - Municipal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council, Dnipro
  - Ivano-Frankivsk National Medical University, Ivano-Frankivsk
  - MNPE "Prykarpatski Clinical Oncological Center" of Ivano-Frankivsk Regional Council", Ivano-Frankivsk
  - Communal enterprise "Kryvyi Rih Oncology Dispensary" of Dnipropetrovsk Regional Council, Kryvyi Rih
- United Kingdom (6):
  - Freeman Hospital, Newcastle upon Tyne, HIGH Heaton
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Heartlands Hospital, Birmingham
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - Hammersmith Hospital, London
  - Churchill Hospital - Oncology, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kopetz S, Tabernero J, Elez E. BREAKWATER Phase III: results for encorafenib and cetuximab plus mFOLFOX6 in first-line BRAF V600E-mutant metastatic colorectal cancer. Future Oncol. 2025 Dec;21(28):3585-3588. doi: 10.1080/14796694.2025.2579882. Epub 2025 Nov 13. PMID 41230651
- [Derived] Elez E, Yoshino T, Shen L, Lonardi S, Van Cutsem E, Eng C, Kim TW, Wasan HS, Desai J, Ciardiello F, Yaeger R, Maughan TS, Morris VK, Wu C, Usari T, Laliberte R, Dychter SS, Zhang X, Tabernero J, Kopetz S; BREAKWATER Trial Investigators. Encorafenib, Cetuximab, and mFOLFOX6 in BRAF-Mutated Colorectal Cancer. N Engl J Med. 2025 Jun 26;392(24):2425-2437. doi: 10.1056/NEJMoa2501912. Epub 2025 May 30. PMID 40444708
- [Derived] Kopetz S, Yoshino T, Van Cutsem E, Eng C, Kim TW, Wasan HS, Desai J, Ciardiello F, Yaeger R, Maughan TS, Beyzarov E, Zhang X, Ferrier G, Zhang X, Tabernero J. Encorafenib, cetuximab and chemotherapy in BRAF-mutant colorectal cancer: a randomized phase 3 trial. Nat Med. 2025 Mar;31(3):901-908. doi: 10.1038/s41591-024-03443-3. Epub 2025 Jan 25. PMID 39863775
- [Derived] Van Cutsem E, Taieb J, Yaeger R, Yoshino T, Grothey A, Maiello E, Elez E, Dekervel J, Ross P, Ruiz-Casado A, Graham J, Kato T, Ruffinelli JC, Andre T, Carriere Roussel E, Klauck I, Groc M, Vedovato JC, Tabernero J. ANCHOR CRC: Results From a Single-Arm, Phase II Study of Encorafenib Plus Binimetinib and Cetuximab in Previously Untreated BRAFV600E-Mutant Metastatic Colorectal Cancer. J Clin Oncol. 2023 May 10;41(14):2628-2637. doi: 10.1200/JCO.22.01693. Epub 2023 Feb 10. PMID 36763936
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4221015